CLINICAL TRIAL: NCT06558812
Title: Evaluation of the Success Rate of Prefabricated Versus Conventional Band and Loop Space Maintainers in Children With Prematurely Lost First Primary Molars A Randomized Clinical Trial
Brief Title: Evaluation of the Success Rate of Prefabricated Versus Conventional Band and Loop Space Maintainers in Children With Prematurely Lost First Primary Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, amal fathy mahmoud mohammed elsayed saker, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Prefabricated space maintainer
Record Dates: First submitted 2024-08-12; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Premature Tooth Exfoliation

STUDY DESIGN:
Intervention Model Description: A randomized controlled clinical trial, parallel group, allocation ratio 1:1 Framework superiority
Who Masked: Outcomes Assessor
Masking Description: Blinding will not be feasible neither for the operator nor the patient. As there are some differences in the clinical steps, the form of the appliances and number of needed visits.
  Outcome assessor and Statistician will be blinded from the intervention and control not knowing which group represents which procedure.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional space maintainer (Other): Conventional band and loops have been widely used with a high rate of success as the most practical way of space maintenance, as reported in numerous articles . Band and loop space maintainer is used to maintain space for successors of early lost primary molars. This is due to the ease and practicality of fabrication, adjustments and repairs of this space maintainer, as well as its ability to continue to function until the eruption of the permanent successor without interfering with their eruption The need for at least two visits to delivery, therefore cannot be planned in patients under general anesthesia. Fabrication of conventional and loop requires an alginate impression and laboratory work.
  Interventions: Device: conventional space maintainer
- prefabricated space maintainer (Other): Prefabricated band and loop devices have been introduced to dentistry in recent times. They can possibly overcome most of the previously mentioned limitations of conventional space maintainers. The prefabricated band and loop space maintainer is adjusted and applied in one visit and therefore can be planned in patients under general anesthesia. Other advantages include less time, more patient and parent satisfaction, and no laboratory work
  Interventions: Device: prefabricated space maintainer

INTERVENTIONS:
Device: prefabricated space maintainer — i. Prefabricated band will be selected for the abutment tooth by measuring the mesiodistal diameter of the abutment tooth with a caliper and will be adjusted with the internal diameter of the prefabricated band.
  ii. The loop will be selected based on the available mesiodistal space and buccolingual width of the abutment tooth, excessive length with be cut by cutting plier and will then place inside the band's tube by using a HOWE pliers.
  iii. Cotton roll isolation will use, then will be cemented with glass ionomer,
  Other Names: chair side space maintainer
  Arms: prefabricated space maintainer
Device: conventional space maintainer — i. A full arch Impressions will be taken with alginate material. ii. Impressions will be poured up using dental stone within 30 min of the impression taking.
  iii. The children will be given an appointment for space maintainer insertion. iv. In the second visit , Cotton roll isolation will use, cementation will be performed with glass ionomer .
  Arms: conventional space maintainer

SUMMARY:
To assess the clinical efficacy of prefabricated space maintainers compared to conventional ones, focusing on preserving the integrity of each component of bands and loops, avoidance of soft tissue impingement as well as preservation of arch dimensions.

DETAILED DESCRIPTION:
Management of the developing occlusion lies firmly within the scope of pediatric dentistry, therefore protection of dental arch integrity and inter-arch relations in the premature loss of teeth can be guaranteed by placing space maintainers. Conventional appliances are used successfully as space maintainers, although they have some disadvantages.The need for at least two visits to delivery, therefore cannot be planned in patients under general anesthesia. Fabrication of conventional and loop requires an alginate impression and laboratory work.

Prefabricated band and loop devices have been introduced to dentistry in recent times. They can possibly overcome most of the previously mentioned limitations of conventional space maintainers. The prefabricated band and loop space maintainer is adjusted and applied in one visit and therefore can be planned in patients under general anesthesia. Other advantages include less time, more patient and parent satisfaction, and no laboratory work

ELIGIBILITY:
Inclusion Criteria:

* Clinical criteria Medically free children.

  * Patient and parent showing cooperation and compliance.
  * Patients having mandibular first deciduous molar indicated for extraction due to extensive coronal caries beyond possible repair, root caries and/or failed pulp therapy.
  * Freshly extracted single molars unilaterally or bilaterally
  * Unilateral or bilateral loss of primary molars before or after the eruption of the first permanent molar
  * Caries free or restored the mandibular second primary molars and deciduous canines in the side of the extraction maintained throughout the entire follow-up period.

Radiographic criteria

* Presence of succedaneous tooth bud.
* Presence of at least 1 mm bone overlying the succedaneous tooth germ
* 1/3 to less than 2/3 of the root of the permanent successor is formed to the prematurely lost primary molars.

Exclusion Criteria:

* • Children with any parafunctional habits.

  * Children with previous allergies to stainless steel.
  * Permanent successors with 2/3 of its roots formed and space analysis does not indicate the fabrication of space maintainer.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
appliance success | 0-3-9 month
  evaluation of clinical success criteria ( • Integrity of each component of band and loop - solder breakdown - decementation - abutment fracture - Soft tissue impingement ) Clinical examination by operator ( binary yes or no )

SECONDARY OUTCOMES:
Space loss between the abutment teeth. | 0-9 month
  • Change in distance measured on digital cast between the mesial midpoint of the second deciduous molar and the distal midpoint of the primary canine in mm
arch dimension | 0-9 month
  measured each of
  1. Arch perimeter by measured on a digital cast as a sum of the incisor, canine and molar segment width in mm
  2. Inter canine width = Measured on a digital cast from cusp tip of canine on one side to cusp tip of canine on the other side in mm
  3. Intermolar width = Measured on a digital cast from central fossa of the second primary molar on one side to central fossa of the second primary molar on the other side in mm
• Patient satisfaction | during insertion of appliance
  Patient-reported using 5-point Likert-type scale from 1-5 face scale
• Cost effectiveness | through study completion , an average of 9 month
  Manually by incremental effectiveness cost ratio ,measuring unit is financial units per result

CONTACTS AND LOCATIONS:
Overall Officials: Dina Yousry El Kharadly, Lecturer, Study Director — October 6 University

REFERENCES:
- [Background] Tahririan D, Safaripour M, Eshghi A, Bonyadian AH. Comparison of the longevity of prefabricated and conventional band and loops in children's primary teeth. Dent Res J (Isfahan). 2019 Nov 12;16(6):428-434. eCollection 2019 Nov-Dec. PMID 31803390
- [Background] Tyagi M, Rana V, Srivastava N, Kaushik N, Moirangthem E, Gaur V. Comparison of the Conventional Band and Loop Space Maintainers with Modified Space Maintainers: A Split-mouth Randomized Clinical Trial. Int J Clin Pediatr Dent. 2021;14(Suppl 1):S63-S68. doi: 10.5005/jp-journals-10005-2046. PMID 35082470
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31803390/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35082470/